CLINICAL TRIAL: NCT05560594
Title: Explorative Study Investigating the Urinary Bladder and Prostate During Intermittent Catheterization in Healthy Male Adults by Use of MR-scanning.
Brief Title: Investigate Bladder and Prostate During Emptying With Intermittent Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP336
Record Dates: First submitted 2022-08-02; First posted 2022-09-29 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Urinary Function

STUDY DESIGN:
Intervention Model Description: Explore the behavior of the urinary bladder and prostate during emptying the bladder with an intermittent catheter.
  By use of 3D scanning techniques and dynamic MRI, the objective is to investigate behavior of bladder emptying using an intermittent catheter compared to the voluntary bladder emptying.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent catheter (Other): Coloplast SpeediCath CH12 male intermittent catheter
  Interventions: Device: Coloplast SpeediCath CH12 standard male intermittent catheter

INTERVENTIONS:
Device: Coloplast SpeediCath CH12 standard male intermittent catheter — Drainage of the bladder through the urethra when using the SpeediCath standard male intermittent catheter.

SUMMARY:
Explorative study investigating the urinary bladder and prostate during intermittent catheterization in healthy male adults by use of MR-scanning.

DETAILED DESCRIPTION:
12 healthy male adults will be enrolled in the investigation. The study includes one study visit where MR-scans of the bladder and prostate will be performed during normal voiding as baseline measurement followed by measurements during emptying of the bladder with an intermittent catheter (SpeediCath CH12 standard male intermittent catheter).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Has given written informed consent
* Be at least 18 years of age and have full legal capacity

Exclusion Criteria:

* Participate in any other clinical investigation
* Has symptoms of UTI (Investigator's judgement)
* Has known abnormalities and/or diseases in the bladder and/ or the lower urinary tract
* Has had previous disease or surgery in lower urinary tract
* Has any MR-scanning contraindication - according to "MR check list"

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male adults
Enrollment: 12 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Bladder morphology | Within 1 year after termination
  Evaluate bladder morphology and behavior during emptying of the bladder by performance of 3D and dynamic MRI
Bladder behavior | Within 1 year after termination
  Evaluate bladder behavior when emptying the bladder with an intermittent catheter evaluated by performance of 3D and dynamic MRI

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, PI, Principal Investigator — Per.bagi@regionh.dk /+45 35 45 83 10
Locations (1):
- Rigshospitalet, Copenhagen, Denmark